CLINICAL TRIAL: NCT01779180
Title: The Effect of Vitamin A Supplementation at Birth on the Development of Atopy in Childhood: Long-term Follow-up of a Randomised Placebo-controlled Trial
Brief Title: Vitamin A Supplementation at Birth and Atopy in Childhood
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bandim Health Project (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-VAS-Atopy
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-02

CONDITIONS: Atopy; Asthma; Eczema; Food Allergy
Keywords: Vitamin A supplementation; BCG vaccination; diphtheria-tetanus-pertussis vaccination; measles vaccination; atopy
MeSH Terms: conditions — Asthma; Eczema; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
INTRODUCTION Eight trials studying the effect of providing neonatal vitamin A supplementation (NVAS) have been reported, and another four are underway to test whether NVAS should become WHO policy. Three of the four African trials were conducted by the Bandim Health Project (BHP) in Guinea-Bissau. One of them was a two-by-two factorial trial among low-birth-weight children. From 2004-2008, the children were randomly allocated to 25,000 IU vitamin A or placebo at birth, and furthermore to BCG vaccination at birth or later as is local policy. In 2011, the investigators conducted a follow-up study. A remarkably strong harmful effect of NVAS on atopy and wheezing was found (manuscript under review).

Seen in the context that NVAS may soon become a WHO policy it is obviously worrying if NVAS is associated with a higher risk of atopy and wheezing. The investigators therefore aim to conduct a similar follow-up study of participants in the first NVAS trial conducted in Guinea-Bissau from 2002-2004, among normal-birth-weight infants, to test whether NVAS is associated with an increased risk of atopy and wheezing and other allergic symptoms as well as growth.

METHODS

Study population:

From 2002-2004 BHP conducted a randomised trial of NVAS. The investigators recruited newborns when they came for BCG vaccination. Provided parental consent, they received an oral supplement of 50,000 IU vitamin A or placebo.

Study design:

This study will be a follow-up study of the cohort of children randomised to NVAS (intervention) or placebo (current policy) together with BCG vaccine at birth.

Other exposures:

The investigators will also investigate the effect of receiving an additional dose of measles vaccine and the timing of DTP vaccine on the development of atopy.

Assessment of outcomes:

The investigators will visit all children at the last known address. Height, weight and mid upper arm circumference will be measured. BCG scar will be examined and vaccination card details recorded by the field assistant. Children will be excluded from skin prick testing (SPT) if they have a history suggestive of anaphylaxis or are currently using anti-histamine medication. SPT will be performed using aero-allergens, food allergens and positive histamine and negative saline control. The mother or guardian will be interviewed by a local assistant. Symptoms of eczema and asthma as well as food allergy will be assessed.

Statistical analysis:

Effect of randomisation group and other factors on outcomes will be analysed in multivariable regression models. All analyses will be adjusted for skin prick tester. All analyses will be conducted stratified by sex.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at birth in NCT00168610

Exclusion Criteria:

* Children with history suggestive of anaphylaxis will be excluded from skin prick testing but included in the study population

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants in a previous neonatal vitamin A supplementation trial
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Atopic sensitisation | Single observation on day of recruitment
  Skin prick test positivity. A wheal >=3mm will be considered positive.

SECONDARY OUTCOMES:
Symptoms of asthma | Single observation on day of recruitment
  Questionnaire based on ISAAC survey for 6-7 year olds
Symptoms of eczema | Single observation on day of recruitment
  Questionnaire based on ISAAC survey for 6-7 year olds
Symptoms of food allergy | Single observation of day of recruitment
  Questionnaire based on Health Nuts survey

OTHER OUTCOMES:
Weight | Single observation on day of recruitment
Height | Single observation on day of recruitment
Mid-upper arm circumference | Single observation on day of recruitment
Hospitalisations | Single observation on day of recruitment
Infectious diseases | Single observation on day of recruitment
  History of chickenpox or measles

CONTACTS AND LOCATIONS:
Overall Officials: Christine Benn, DMSc, Principal Investigator — Statens Serum Institut
Locations (1):
- Bandim Health Project, Bissau, Bissau Codex, Guinea-Bissau

REFERENCES:
- [Derived] Aage S, Kiraly N, Da Costa K, Byberg S, Bjerregaard-Andersen M, Fisker AB, Aaby P, Benn CS. Neonatal vitamin A supplementation associated with increased atopy in girls. Allergy. 2015 Aug;70(8):985-94. doi: 10.1111/all.12641. Epub 2015 May 18. PMID 25939706